CLINICAL TRIAL: NCT00955903
Title: Calorie Restriction and Changes in Body Composition, Disease, Function, and Quality of Life in Older Adults
Acronym: CROSSROADS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jamy Ard, MD, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: F090430012
Record Dates: First submitted 2009-08-06; First posted 2009-08-10 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Obesity; Diabetes; Hypertension; Hyperlipidemia
Keywords: glucose; insulin; lipids; C-reactive protein; adiponectin; leptin; TNF alpha; IL-6; Quality of Life; functional status
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Hypertension; Hyperlipidemias; Insulin Resistance | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Weight Loss (Experimental): Participants receive Exercise and Reduced Calorie Diet Interventions
  Interventions: Behavioral: Exercise; Behavioral: Reduced Calorie Diet
- Control (Active Comparator): Participants receive Exercise Intervention
  Interventions: Behavioral: Exercise
- Weight Maintenance (Active Comparator): Participants receive Exercise and a Weight Maintenance Diet Interventions
  Interventions: Behavioral: Exercise; Behavioral: Weight Maintenance Diet

INTERVENTIONS:
Behavioral: Exercise — Participants will participate in supervised exercise sessions
Behavioral: Reduced Calorie Diet — Participants will follow a reduced calorie diet
  Arms: Weight Loss
Behavioral: Weight Maintenance Diet — Participants will follow a weight maintenance diet
  Arms: Weight Maintenance

SUMMARY:
The investigators want to determine if the benefits of weight loss outweigh the potential risk in a group of older adults. The investigators will test the hypothesis that changes in diet composition alone or in conjunction with weight loss will have a significant effect on fat stores, and as a result, improve cardiometabolic risk factors and functional status in adults 65 and older.

ELIGIBILITY:
Inclusion Criteria:

* at least 65 years of age
* BMI 27 - 42 kg/m2 - at increased health risk (taking at least 1 medication for hypertension, hyperlipidemia, or type 2 diabetes)

Exclusion Criteria:

* difficulties chewing or swallowing food
* digestive diseases that may affect the ability to follow a high fiber diet
* cognitive impairment
* depression
* recent weight change (+/- 10 lbs in the last 12 months)
* poorly controlled blood pressure
* history of non-skin cancer in last 5 years
* cardiovascular disease event in past 6 months or severe pulmonary disease or renal failure
* major liver dysfunction
* current smoker or quit less than months prior
* history of prior surgical procedures for weight control or liposuction
* use of estrogen or testosterone replacement therapy
* current use of insulin or sulfonylurea agents
* current use of corticosteroids > 5 days/month on average
* current use of medications for treatment of psychosis or manic-depressive illness
* use of weight-loss medications in previous 3 months
* dependence on others for food procurement or preparation
* ischemic changes on exercise treadmill test

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 167 (Actual)
Dates: Start 2010-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamy D Ard, MD, Principal Investigator — University of Alabama at Birmingham; Julie Locher, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Senkus KE, Crowe-White KM, Bolland AC, Locher JL, Ard JD. Changes in adiponectin:leptin ratio among older adults with obesity following a 12-month exercise and diet intervention. Nutr Diabetes. 2022 Jun 2;12(1):30. doi: 10.1038/s41387-022-00207-1. PMID 35654771
- [Derived] Senkus KE, Crowe-White KM, Locher JL, Ard JD. Relative fat mass assessment estimates changes in adiposity among female older adults with obesity after a 12-month exercise and diet intervention. Ann Med. 2022 Dec;54(1):1160-1166. doi: 10.1080/07853890.2022.2067352. PMID 35471192
- [Derived] Bragg AE, Crowe-White KM, Ellis AC, Studer M, Phillips F, Samsel S, Parton J, Locher JL, Ard JD. Changes in Cardiometabolic Risk Among Older Adults with Obesity: An Ancillary Analysis of a Randomized Controlled Trial Investigating Exercise Plus Weight Maintenance and Exercise Plus Intentional Weight Loss by Caloric Restriction. J Acad Nutr Diet. 2022 Feb;122(2):354-362. doi: 10.1016/j.jand.2021.07.009. Epub 2021 Sep 1. PMID 34486528
- [Derived] Crowe-White KM, Ellis AC, Mehta T, Locher JL, Ard JD. Dietary Quality Assessed by the HEI-2010 and Biomarkers of Cardiometabolic Disease: An Exploratory Analysis. J Am Coll Nutr. 2019 Sep-Oct;38(7):640-647. doi: 10.1080/07315724.2019.1580168. Epub 2019 May 30. PMID 31145045

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 participants were subsequently diagnosed with cancer after enrollment and thus disqualified from continuing in the trial. They were dropped from the analysis.
Groups:
- Weight Loss: Participants receive Exercise Only and Reduced Calorie Diet Interventions
  Exercise Only: Participants will participate in supervised exercise sessions
  Reduced Calorie Diet: Participants will follow a reduced calorie diet
- Control: Participants receive Exercise Only Intervention
  Exercise Only: Participants will participate in supervised exercise sessions
- Weight Maintenance: Participants receive Exercise Only and a Weight Maintenance Diet Interventions
  Exercise Only: Participants will participate in supervised exercise sessions
  Weight Maintenance Diet: Participants will follow a weight maintenance diet
Period: Overall Study
Arm/Group | Weight Loss | Control | Weight Maintenance
Started | 55 | 54 | 55
Completed | 49 | 51 | 48
Not Completed | 6 | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Weight Loss | Control | Weight Maintenance | Total
Number analyzed (Participants) | 55 | 54 | 55 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (4.8) | 69.9 (4.5) | 70.5 (4.8) | 70.3 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 37 | 33 | 102
  Male | 23 | 17 | 22 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 15 | 12 | 39
  White | 42 | 39 | 43 | 124
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 55 | 54 | 55 | 164

OUTCOME MEASURES:

1. Primary Outcome: Change in Abdominal Fat Mass
Description: Visceral adipose tissue (cm3) by MRI. Change is calculated as value at baseline minus value at 1 year
Time Frame: Baseline to 1 year
Measure: Mean (Standard Deviation); unit: Cubic cm
Arm/Group | Weight Loss | Control | Weight Maintenance
Number analyzed (Participants) | 55 | 54 | 55
Cubic cm | -192.6 (185.2) | -21.9 (173.7) | -275 (189.2)

2. Secondary Outcome: Cardiometabolic Risk Factors
Description: We are reporting change in blood glucose. Change is calculated as value at baseline minus value at 1 year
Time Frame: Baseline to 1 year
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Weight Loss | Control | Weight Maintenance
Number analyzed (Participants) | 55 | 54 | 55
mg/dL | -7.2 (2.8) | 1.2 (2.5) | -1.2 (2.5)

3. Secondary Outcome: Weight Change/Maintenance
Description: The change in body weight at follow up of 1 year. Change is calculated as value at baseline minus value at 1 year
Time Frame: Baseline to 1 year
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Weight Loss | Control | Weight Maintenance
Number analyzed (Participants) | 55 | 54 | 55
Kg | -3.9 (0.7) | -1.3 (0.7) | -0.9 (0.7)

ADVERSE EVENTS:
Arm/Group | Weight Loss | Control | Weight Maintenance
Serious Adverse Events (participants affected / at risk) | 8/55 | 11/54 | 12/55
Other Adverse Events (participants affected / at risk) | 36/55 | 36/54 | 40/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weight Loss (N=55) | Control (N=54) | Weight Maintenance (N=55)
Joint surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1)
Chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary symptoms (Renal and urinary disorders) | 0 (0) | 3 (3) | 1 (1)
Heart rate and blood pressure abnormalities (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Complications related to surgery (Surgical and medical procedures) | 1 (1) | 1 (1) | 3 (3)
Pain (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Broken bone (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 2 (2)
Vaginal bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weight Loss (N=55) | Control (N=54) | Weight Maintenance (N=55)
Cardiovascular (Cardiac disorders) | 8 (8) | 14 (14) | 10 (10)
Gastrointestinal (Gastrointestinal disorders) | 12 (12) | 6 (6) | 12 (12)
General, Constitutional (General disorders) | 4 (4) | 3 (3) | 9 (9)
Genitourinary (Renal and urinary disorders) | 1 (1) | 5 (5) | 3 (3)
Muscle and bone issues (Musculoskeletal and connective tissue disorders) | 34 (34) | 35 (35) | 35 (35)
Nervous system (Nervous system disorders) | 8 (8) | 7 (7) | 7 (7)
Psychiatric and mood changes (Psychiatric disorders) | 5 (5) | 4 (4) | 4 (4)

LIMITATIONS AND CAVEATS:
This trial was completed in older adults (age 65+) with at least one major risk factor for heart disease.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No